CLINICAL TRIAL: NCT05339815
Title: Clinical and Radiographic Outcomes of Reverse Shoulder Arthroplasty Performed With 36-mm CoCrMo vs 40-mm Cross-linked UHMWPE Glenospheres.
Brief Title: S-33 SMR Shoulder HP Reverse Glenosphere
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: S-33
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-04

CONDITIONS: Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 36 mm CoCrMo glenospheres
  Interventions: Device: SMR shoulder arthroplasty
- 40 mm cross-linked UHMWPE glenospheres
  Interventions: Device: SMR shoulder arthroplasty

INTERVENTIONS:
Device: SMR shoulder arthroplasty — Data collection of population that underwent a reverse shoulder arthroplasty performed with SMR 36-mm CoCrMo versus 40-mm cross-linked UHMWPE glenospheres

SUMMARY:
Study Design: Single arm, retrospective and prospective, single center, post-market clinical study Purpose:To demonstrate the safety and effectiveness of the SMR Reverse HP Shoulder System device for primary, fracture or revision total shoulder replacement out to 24 months. The eligible study population is the entire population that underwent a reverse shoulder arthroplasty performed with 36-mm CoCrMo versus 40-mm cross-linked UHMWPE glenospheres between January 1, 2013 and January 1, 2020 at Wrightington Hospital (UK) in accordance with the indication for use of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was treated with the SMR Reverse Shoulder System device (either with 36-mm CoCrMo glenosphere or 40-mm cross-linked UHMWPE glenosphere) between January 1, 2013 and January 1, 2020 as per Instruction for Use
2. Patient was an adult male or female and was 18 years of age or older at the time of surgery
3. Patient received the SMR Reverse Shoulder System for primary, fracture, or revision total shoulder replacement in a grossly rotator cuff deficient joint with severe arthroplasty
4. The patient's joint was anatomically and structurally suited to receive the selected implants, with a functional deltoid muscle
5. Surgery date is at least 24 months from screening of data
6. Patient has baseline radiographs and Oxford Shoulder Score

Exclusion Criteria:

1 Patient was treated with the SMR Reverse Shoulder System device (either with 36-mm CoCrMo glenosphere or 40-mm cross-linked UHMWPE glenosphere) between January 1, 2013 and January 1, 2020 out of the Indications for Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible study population is the entire population that underwent a reverse shoulder arthroplasty performed with 36-mm CoCrMo versus 40-mm cross-linked UHMWPE glenospheres between January 1, 2013 and January 1, 2020 at Wrightington Hospital (UK) in accordance with the indication for use of the product.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is based upon achieving composite clinical success (CCS) | From baseline to FU 24 months
  The primary endpoint is based upon achieving composite clinical success (CCS) from baseline to 24-month follow-up measured as:
  - No continuous radiolucent line around the implant
  Glenoid Component Radiolucency will be graded in accordance with the following definitions:
  0. Absent: No evidence of radiolucency > 2 mm in width along the bone-implant interface in any zone.
  1. Present: Presence of radiolucency > 2 mm in width along the bone-implant interface in one or more zones
The primary endpoint is based upon achieving composite clinical success (CCS) | From baseline to FU 24 months
  The primary endpoint is based upon achieving composite clinical success (CCS) from baseline to 24-month follow-up measured as:
  - Change from baseline of the Oxford Should Score ≥ 6 points.
  Oxford Shoulder Score (OSS) is a 12-item patient-reported PRO specifically designed and developed for assessing outcomes of shoulder surgery.
The primary endpoint is based upon achieving composite clinical success (CCS) | From baseline to FU 24 months
  The primary endpoint is based upon achieving composite clinical success (CCS) from baseline to 24-month follow-up measured as:
  - No revision or removals.
  A removal of the glenosphere component is intended as a revision and of the implant.
The primary endpoint is based upon achieving composite clinical success (CCS) | From baseline to FU 24 months
  The primary endpoint is based upon achieving composite clinical success (CCS) from baseline to 24-month follow-up measured as:
  No system-related SAE (device-related)
  Device Related Adverse Events/Serious Adverse Events, device deficiencies, malfunctions and use errors at all follow-up time points.

SECONDARY OUTCOMES:
Assessment of the clinical evaluation of the SMR Reverse glenosphere used in real life settings over a period of 2 years (24 months) through PROMs when available and medical evaluation. | From baseline to FU 24 months
  Measure Oxford shoulder score
  Oxford Shoulder Score (OSS) is a 12-item patient-reported PRO specifically designed and developed for assessing outcomes of shoulder surgery.
Assessment of the clinical evaluation of the SMR Reverse glenosphere used in real life settings over a period of 2 years (24 months) through PROMs when available and medical evaluation. | From baseline to FU 24 months
  Measure Constant Score
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The higher the score, the higher the quality of the function.
Assessment of the clinical evaluation of the SMR Reverse glenosphere used in real life settings over a period of 2 years (24 months) through PROMs when available and medical evaluation. | From baseline to FU 24 months
  Measure American Shoulder and Elbow Surgeons Shoulder Score (ASES)
  American Shoulder and Elbow Surgeons (ASES) score contains a patient self-report section and a section used by medical professionals to record physical examination findings to assess patients with shoulder pathologies.
  The patient self-report section of the ASES is a condition specific scale is intended to measure functional limitations and pain of the shoulder. The pain score is calculated from the single pain question and the function score from the sum of the 10 questions addressing function. The pain score and function composite score are weighted equally (50 points each) and combined for a total score out of a possible 100 points.
  The physician assessment section is composed by 4 parts: motion, stability, strength and physical findings.
Assessment of the clinical evaluation of the SMR Reverse glenosphere used in real life settings over a period of 2 years (24 months) through PROMs when available and medical evaluation. | From baseline to FU 24 months
  Measure Quick DASH
  The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (4 items, scored 1-5). At least 10 of the 11 items must be completed for a score to be calculated. All items are scored on a scale of 5 (Likert) levels: 1 = no difficulty/symptoms, 2 = mild difficulty/symptoms, 3 = moderate difficulty/symptoms, 4 = severe difficulty/symptoms, and 5 = extreme difficulty (unable to do)/symptoms.
  The assigned values for all completed responses are simply summed and averaged, producing a score out of five. This value is then transformed to a score out of 100 by subtracting one and multiplying by 25. This transformation is done to make the score easier to compare to other measures scaled on a 0-100 scale. A higher score indicates greater disability.
Survivorship of the implant (Kaplan-Meier estimate) through 2 years (24 months) of follow-up after surgery | From baseline to FU 24 months
  Kaplan-Meier
Incidence, type and severity of all Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effect (ADEs), Serious Adverse Device Effects (SADEs) | From baseline to FU 24 months
  Device Related Adverse Events/Serious Adverse Events, device deficiencies, malfunctions and use errors at all follow-up time points

CONTACTS AND LOCATIONS:
Locations (1):
- Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan, United Kingdom

IPD SHARING:
Plan to Share IPD: No